CLINICAL TRIAL: NCT07325409
Title: Sports Nutrition Benefits of Weizmannia Coagulans BC99: a Randomized Controlled Trial on Muscle Function and Recovery in Healthy Participants
Brief Title: Sports Nutrition Benefits of Weizmannia Coagulans BC99
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK20251225
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: College Students of the School of Physical Education

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): 3g dose of milk protein concentrate/pack, 8 packs per day
  Interventions: Dietary Supplement: Placebo
- BC99 group (Experimental): 3g dose of milk protein concentrate with 6×109 Colony Forming Unit (CFU) W. coagulans BC99/pack, 8 packs per day
  Interventions: Dietary Supplement: BC99

INTERVENTIONS:
Dietary Supplement: Placebo — The experimental phase of this study lasts 12 weeks and each participant will have 3 visits (week 0, week 6, week 12)
  Arms: Placebo group
Dietary Supplement: BC99 — The experimental phase of this study lasts 12 weeks and each participant will have 3 visits (week 0, week 6, week 12)
  Arms: BC99 group

SUMMARY:
To evaluate the clinical efficacy of Weizmannia coagulans BC99 in young Chinese patients with exercise-induced muscle damage compared with placebo, and to explore its effects on inflammatory responses and intestinal microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 19-35 years, with no restriction on sex;
2. Physically active individuals with regular daily exercise training intensity and duration;
3. No history of allergy to protein products;
4. Body weight ≥50 kg for male subjects and ≥45 kg for female subjects; body mass index (BMI), calculated as weight (kg) divided by height squared (m²), within the range of 19.0-24.0 kg/m²;
5. No history of cardiovascular or cerebrovascular diseases, hypertension, diabetes, hepatic or renal dysfunction, or other underlying diseases or metabolic disorders;
6. Willingness to comply with the study protocol and study restrictions, and voluntary provision of written informed consent to participate in the study.

Exclusion Criteria:

1. History of allergic constitution or immunodeficiency;
2. Blood donation or significant blood loss (≥200 mL) within 3 months prior to administration of the investigational product;
3. Presence of severe diseases of major organs, including the cardiovascular system, lungs, liver, or kidneys, as well as diabetes mellitus, severe thyroid disorders, metabolic diseases, malignant tumors, or severe immune system diseases;
4. Use of medications affecting the intestinal microbiota (including antibiotics, microecological preparations, intestinal mucosal protectants, traditional Chinese medicines, etc.) for more than one consecutive week within 1 month prior to screening;
5. Any other condition that, in the investigator's judgment, makes the subject unsuitable for participation in the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Pain evaluation | 12 weeks
  Visual analog scale (VAS) was used for assessing the pain level of muscle, ranging from 0 to 10 point (0 means no pain; 10 represent worst imaginable pain). VAS scores were recorded at 24h, 48h and 72h after the intense exercise work stress.

SECONDARY OUTCOMES:
Cortisol in plasma | 12 weeks
  This indicator was determined using commercially available assay kits (BYabscience, Nanjing, China).
Peptide YY in plasma | 12 weeks
  This indicator was determined using commercially available assay kits (BYabscience, Nanjing, China).

CONTACTS AND LOCATIONS:
Locations (1):
- Wu Ying, Luoyang, Henan, China